CLINICAL TRIAL: NCT05614622
Title: The Effect of Mydriatics on Posterior Synechia After Combined Surgery of Pars Plana Vitrectomy, Phacoemulsification, and Intraocular Lens Implantation
Brief Title: Mydriatic Drops After Combined Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Yair Pesoa, Dr, Principal Investigator., Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0243-20-RMC
Record Dates: First submitted 2022-10-31; First posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Posterior Synechiae of Iris
MeSH Terms: interventions — Cyclopentolate; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Control group receives standard post-operative treatment, which includes self-instillation of Ofloxacin and Dexamethasone eye drops with tapering down from q.i.d for the 1st week to once daily in the 4th week
- Study (Experimental): The study group receives standard post-operative treatment same as the control group. And additional treatment of a short-acting mydriatic agent (Cyclopentolate Hydrochloride 1.0% eye drops) t.i.d for 4 weeks (to operate eye alone)
  Interventions: Drug: Cyclopentolate Hydrochloride 1.0% eye drops

INTERVENTIONS:
Drug: Cyclopentolate Hydrochloride 1.0% eye drops — A short-acting mydriatic agent
  Arms: Study

SUMMARY:
The study goal is to evaluate the influence of mydriatic drops on the development of posterior synechia after combined cataract and vitrectomy surgery.

DETAILED DESCRIPTION:
Cataract and vitreoretinal disorders often coexist, and with up to 80 percent chance for cataract formation following vitreoretinal surgery within the first year, combined surgery of phacoemulsification, pars plana vitrectomy (PPV) and intraocular lens (IOL) implantation has become increasingly accepted.

The main advantages of combined surgery include better visualization during surgery and the elimination of the need for additional surgery, which translates to overall quicker visual recovery and cost-effectiveness. Like the more exercised, two-step procedure, the combined surgery was shown to be safe and effective with relatively few complications. However, one complication seen more frequently after the combined surgery is postoperative anterior chamber inflammatory response, and with it, the formation of posterior synechia, reaching an average of 18 percent.

The development of posterior synechia interferes with postoperative visualization of the fundus, thus diminishing an important advantage of the combined procedure. Moreover, in a few cases, it can even be complicated by angle closure glaucoma.

Currently, there is no consensus on whether postoperative treatment after combined surgery should include additional treatment to help prevent the formation of synechia. The frequency and severity of posterior synechia after a combined operation may be reduced using short-acting mydriatics. However, there is no sufficient data nor a prospective study to support this as common practice. It is, therefore, we sought to better evaluate the effect of topical short-acting mydriatics on the formation of posterior synechia after combined surgery and compare it with standard postoperative treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent combined cataract and vitrectomy surgery with IOL implantation.

Exclusion Criteria:

* History of uveitis prior to surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-11-10 (Actual); Primary Completion 2022-01-03 (Actual); Study Completion 2022-01-03 (Actual)

PRIMARY OUTCOMES:
Number of participants developed iris posterior synechiae after surgery | 24 weeks
  Iris posterior synechia is an adhesion formed between the iris and the capsular bag, which holds the implanted lens in place. It is a relatively common complication observed after intra-ocular surgery. Viewed under the slit lamp at the standard ophthalmologist examination after surgery.
  Mild to Moderate synechia can interrupt pupil dilatation and interfere with postoperative visualization of the fundus, thus diminishing an advantage of the combined surgery.
  Substantial synechia may affect the movement of the aqueous from the posterior to the anterior chamber resulting in secondary angle closure glaucoma.

CONTACTS AND LOCATIONS:
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: Undecided